CLINICAL TRIAL: NCT01519141
Title: Immunologic and Inflammatory Factors and Cardiovascular Risk in Patients With HIV Infection or Autoimmune Diseases
Brief Title: Inflammation, Viral Replication, and Atherosclerosis in Treated HIV Infection
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01HL095130 (NIH); 5R01HL095130 (NIH)
Record Dates: First submitted 2012-01-12; First posted 2012-01-26 (Estimated); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Atherosclerosis
Keywords: Human Immunodeficiency Virus; Atherosclerosis; Inflammation; Endothelial Function; Thrombosis
MeSH Terms: conditions — Atherosclerosis; Acquired Immunodeficiency Syndrome; Inflammation; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV-negative controls: HIV-negative individuals
- HIV-infected patients: HIV-infected patients who are on a stable antiretroviral drug regimen for at least a year; all plasma HIV RNA levels within the past year must be below conventional levels of detection (< 50 copies RNA/mL).

SUMMARY:
This is a longitudinal observational study of HIV-infected patients and HIV-negative control patients that is being conducted to learn more about immunologic factors, inflammation, and cardiovascular risk in patients with HIV infection or in patients with autoimmune disease. The investigators plan to obtain measurement of carotid artery intima media thickness (IMT) using high resolution ultrasound as a noninvasive means for tracking atherosclerotic progression. The investigators will also measure lipid and lipoprotein levels, inflammatory markers, markers of Cytomegalovirus (CMV) infection, thrombotic markers, atherogenic lipoproteins, and markers of immune function. Immunophenotyping will be performed on freshly collected blood and analyzed by flow cytometry to identify activated T-cells, T-cell turnover, proportions of T-cells, and CMV function. HIV-infected patients will have CD4 count and HIV viral load measured in addition. Patients will undergo detailed clinical history including HIV disease, specific HIV medications, comorbid conditions, and health related behaviors. Physical exam and measurements will be obtained to assess for the presence of lipodystrophy. Patients will undergo study visits for ultrasound, blood draw, and interview at 4-12 month intervals for the next 3 years.

Patients will also go assessment of endothelial function, endothelial progenitor cells, arterial stiffness as measured using pulse wave tonometry.

To demonstrate the feasibility of a larger scale investigation of cardiac arrhythmia in HIV positive and negative patients with cardiac disease, the investigators will use 48-hour Holter monitor surveillance to monitor HIV-infected and uninfected patients with a history of myocardial infarction, systolic left ventricular dysfunction, and/or pulmonary artery hypertension for the presence of cardiac arrhythmia.

The FDG PET scan (18F-fluorodeoxyglucose positron emission tomography-computed tomography) will be used to detect and quantify inflammation in the body.

DETAILED DESCRIPTION:
This proposal is currently approved by CHR (#H9577-18534-03C, exp date 3/26/04); the purpose of this new application is to split the currently approved protocol into a separate protocol with a separate PI. Data collected and patients seen under the previously approved protocol will be carried over into this new separate protocol. This is a longitudinal observational study of HIV-infected patients and HIV-negative control patients, and individuals with autoimmune diseases. We plan to obtain measurement of carotid artery intima media thickness (IMT) using high resolution ultrasound as a noninvasive means for tracking atherosclerotic progression. In addition, patients will undergo ct scan for coronary calcium and single slice abdominal ct scan to assess visceral fat. We will also measure lipid and lipoprotein levels, inflammatory markers, markers of CMV infection, thrombotic markers, atherogenic lipoproteins, and markers of immune function. Immunophenotyping will be performed on freshly collected blood and analyzed by flow cytometry to identify activated T cells,T cell turnover, proportions of T cells, and CMV function. HIV-infected patients will have CD4 count and HIV viral load measured in addition. Patients will undergo detailed clinical history including HIV disease, specific HIV medications, comorbid conditions, and health related behaviours. Physical exam and measurements will be obtained to assess for the presence of lipodystrophy. Patients will undergo study visits for ultrasound, blood draw, and interview at 4-12 month intervals for the next 3 years. Patients will also go assessment of endothelial function, endothelial progenitor cells, arterial stiffness as measured using pulse wave tonometry. In patients with detectable calcium on CT scan, they will be given the option of obtaining CT angiography. Patients will also undergo testing for peripheral arterial disease using ankle brachial index testing and exercise treadmill testing.

ELIGIBILITY:
Inclusion Criteria:

* Stable antiretroviral therapy for at least 12 months, and have no immediate plans to alter therapy.
* All plasma HIV RNA levels within the past year must be below conventional levels of detection (< 50 copies RNA/mL), although isolated single values > 50 but < 1000 copies will be allowed if they were preceded and followed by undetectable viral load determinations.
* Ability to provide reliable history of HIV medications or has received the majority of medical care from San Francisco General Hospital with available records of medical treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 325 well-characterized HIV-infected individuals and 75 HIV-uninfected individuals.
Sampling Method: Non-Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2003-07; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
carotid intima-media thickness | 2 years
  Increased carotid intima-media thickness (mm)
brachial artery flow-mediated dilatation | 2 years
  decreased brachial artery flow-mediated dilatation (%)
D-dimer | 2 years
  Increased D-dimer levels (mcg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Hsue, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Hsue PY, Scherzer R, Hunt PW, Schnell A, Bolger AF, Kalapus SC, Maka K, Martin JN, Ganz P, Deeks SG. Carotid Intima-Media Thickness Progression in HIV-Infected Adults Occurs Preferentially at the Carotid Bifurcation and Is Predicted by Inflammation. J Am Heart Assoc. 2012 Apr;1(2):jah3-e000422. doi: 10.1161/JAHA.111.000422. Epub 2012 Apr 24. PMID 23130122